CLINICAL TRIAL: NCT05124236
Title: A Multicenter Prospective, Interventional, Randomized Trial of Preoperative Radiosurgery Compared with Postoperative Stereotactic Radiotherapy for Resectable Brain Metastases
Brief Title: Trial of Preoperative Radiosurgery Versus Postoperative Stereotactic Radiotherapy for Resectable Brain Metastases
Acronym: PREOP-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Susanne Rogers (Other)
Collaborators: University of Basel (Other)
Responsible Party: Sponsor-Investigator, Susanne Rogers, Sponsor-Investigator, Kantonsspital Aarau
Organization: Kantonsspital Aarau (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 410.000.146
Record Dates: First submitted 2021-10-14; First posted 2021-11-17 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-09

CONDITIONS: Brain Metastases, Adult
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Preoperative radiosurgery (Experimental): The interventional arm is single fraction preoperative radiosurgery to a brain metastasis identified for neurosurgical resection.
  Interventions: Radiation: preoperative radiosurgery
- Postoperative hypofractionated stereotactic radiotherapy (Active Comparator): The active comparator arm is the standard of care of postoperative hypofractionated stereotactic radiotherapy to the surgical cavity in 5 fractions following resection of the brain metastasis.
  Interventions: Radiation: postoperative hypofractionated stereotactic radiotherapy

INTERVENTIONS:
Radiation: preoperative radiosurgery — single fraction radiosurgery
  Arms: Preoperative radiosurgery
Radiation: postoperative hypofractionated stereotactic radiotherapy — 5 fraction stereotactic radiotherapy /fractionated radiosurgery
  Arms: Postoperative hypofractionated stereotactic radiotherapy

SUMMARY:
The research question is whether a single fraction of preoperative radiosurgery can reduce the incidence of leptomeningeal disease 12 months following resection of a brain metastasis (BM) as compared with 5 fractions of postoperative stereotactic radiotherapy.

DETAILED DESCRIPTION:
Neurosurgical resection of a brain metastasis in patients with a diagnosis of cancer may be indicated however the recurrence rate approximates 50% and adjuvant radiotherapy is standard. Single fraction postoperative stereotactic radiosurgery (SRS) has been widely adopted as a standard therapy as it achieves equivalent survival and prevents loss of neurocognitive function as compared with whole brain radiotherapy and improves cavity local control rates as compared with observation. Hypofractionated stereotactic radiotherapy in 3 to 5 fractions (hfSRT) is also used in the postoperative setting.

Nodular leptomeningeal disease (nLMD) is a recognised pattern of failure after postoperative SRS and hfSRT. A 16.9% incidence of nodular LMD was seen after surgery and a similar incidence of 11%-28%is reported following postoperative SRS in retrospective series. These data suggest that postoperative SRS/hfSRT have no significant effect on the development of LMD following surgery.

The incidence of LMD following single fraction preoperative SRS is only 6.1% according to the largest retrospective series. Preoperative SRS takes advantage of the easier delineation of an intact BM and sterilizes tumor cells disseminated at surgery. Side effects are minimized by a smaller planning margin, a dose reduction and resection of the irradiated volume. In addition, there is no delay to systemic therapy due to wound healing/complications. Furthermore, a single fraction offers patient convenience.

This trial will randomise and compare intracranial outcomes between single fraction preoperative SRS and 5 fraction postoperative hFSRT.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Age ≥18
4. Karnofsky performance status ≥60
5. Histological diagnosis of a malignant primary or metastatic tumour
6. Ability to take steroids
7. No contraindication to magnetic resonance imaging (MRI)
8. MRI-diagnosis of a clearly demarcated contrast-enhancing brain metastasis up to 4.0 cm diameter indicated for neurosurgical resection (tumorboard decision). Up to 3 other brain metastases suitable for primary radiosurgery/ stereotactic radiotherapy
9. Survival estimated by primary clinician > 12 months
10. Platelet count > 100/ml, INR < 1.3, Hb > 7.5 g/dL

Exclusion Criteria:

1. Radiosensitive histology: germ cell tumour, lymphoma, multiple myeloma
2. >10 mm midline shift, effacement of the 4th ventricle or other sign of raised intracranial pressure requiring urgent decompressive surgery
3. More than 4 brain metastases or the diameter of the metastasis for resection >4.0 cm.
4. More than 1 metastasis requiring resection
5. Leptomeningeal disease in the CSF or on MRI (unless localized and can be irradiated then resected with the metastasis)
6. Prior radiation to the brain (SRS/SRT to lesion to be resected and /or WBRT)
7. Prior resection of a primary or secondary brain tumor
8. Prior diagnosis of a non-meningioma brain tumor
9. Prior radionuclide therapy within 30 days
10. Prior anti-VEGF therapy within 6 weeks
11. Unable to tolerate radiosurgery immobilization and treatment
12. Inability to give informed consent
13. Pregnancy or lactation
14. Females of reproductive potential not willing to use effective contraception for at least 6 months after radiotherapy
15. Males of reproductive potential not effective contraception for 3 months after radiotherapy
16. Lack of likely compliance with protocol and follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-07-29 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Leptomeningeal disease | 12 months after intervention
  time to Leptomeningeal disease

SECONDARY OUTCOMES:
Local control of the surgical cavity | 12 months after intervention
  No evidence of tumour recurrence on contrsat-enhanced MRI
Distant brain failure | 12 months after intervention
  New brain metastases
Radionecrosis | 12 months after intervention
  Adverse radiation effects
Quality of life assessment | 3,6,12 months after intervention
  EORTC questionnaire core questionnaire QLQ30, EORTC questionnaire brain module BN 20 (1-4, low scores reflect better QoL)

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Rogers, MD PhD, Principal Investigator — Kantonsspital Aarau, Radio-Onkologie-Zentrum Mittelland
Locations (8):
- Tirol Kliniken Innsbruck, Innsbruck, Austria
- Universitätsklinikum Schleswig Holstein, Kiel, Germany
- Switzerland (6):
  - Kantonsspital Aarau, Aarau, Canton of Aargau
  - Inselspital, Universitätsklinik für Radio-Onkologie, Bern, Freiburgstrasse
  - Kantonsspital Graubünden, Chur
  - Luzerner Kantonsspital, Lucerne
  - Kantonsspital St. Gallen, Sankt Gallen
  - Kantonsspital Winterthur, Winterthur

IPD SHARING:
Plan to Share IPD: No